CLINICAL TRIAL: NCT02391467
Title: Validity of Non-invasive Liver Fibrosis Assessment by Ultrasound-based Elastography at the Third Trimester of Pregnancy: a Prospective Study
Brief Title: Validity of Elastography During Pregnancy
Status: Suspended | Type: Observational
Why Stopped: issue concerning safety of elastography during pregnancy
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Stephane Mouly, MD PhD, Professor Paris VII University, Paris, France, Hopital Lariboisière
Other Study IDs: Liver006
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis B Virus Infection; Pregnant Women
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Non invasive methods are the only available methods to stage liver fibrosis during pregnancy. The safety of elastometry - ultrasound based - is obvious, as medical supervision of pregnancy is based on ultrasonography, both methods using same wavelengths. Therefore, this method is sometimes used in pregnant women with recent diagnosis of chronic viral hepatitis infection, whereas its validity in pregnant women has never been studied. This lack of data justifies our study.

DETAILED DESCRIPTION:
One measurement during the third trimester of pregnancy will be compared to a second measurement, 3 months after childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Followed in Obstetrics Dpt
* HBV or HCV chronic hepatitis
* After information and written consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women with HBV or HCV chronic hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Difference between the fibrosis score during and after pregnancy | 3 to 6 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O SELLIER, MD, PhD, Principal Investigator — Hopital Lariboisiere, Paris, France
Locations (1):
- Hopital Lariboisiere, Paris, France